CLINICAL TRIAL: NCT01126099
Title: Prazosin Treatment for Disruptive Agitation in Alzheimer's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Institute for Biomedical and Clinical Research (Other)
Collaborators: National Institute on Aging (NIA) (NIH); VA Puget Sound Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1R01AG033133-01A1 (NIH); 5R01AG033133 (NIH)
Record Dates: First submitted 2010-05-17; First posted 2010-05-19 (Estimated); Results first posted 2015-05-21 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Alzheimer's Disease
Keywords: double-blind; treatment; prazosin; Disruptive behaviors in Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Prazosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prazosin (Experimental): In the double blind phase (12 weeks), study participants will take either prazosin for placebo. For the open label phase (12 weeks), all study participants will take prazosin.
  Interventions: Drug: Prazosin
- Placebo (Placebo Comparator): In the double blind phase (12 weeks), study participants will take either prazosin for placebo. For the open label phase (12 weeks), all study participants will take prazosin.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prazosin — 4 mg capsules twice daily for 12 weeks
  Other Names: minipress
  Arms: Prazosin
Drug: Placebo — Placebo capsules twice daily for 12 weeks
  Other Names: inert substance
  Arms: Placebo

SUMMARY:
A study of outpatient participants with Alzheimer's disease or a related dementia who have difficult behaviors that are upsetting for them or their caregivers. Prazosin is a medication that is commonly used to treat people with high blood pressure. Research with prazosin has shown that it may be effective in treating behavioral problems by reducing excess adrenalin effects in the brain.

DETAILED DESCRIPTION:
This is a 24 week study with 14 visits to the research clinic. Approximately 6 of these visits may be done by phone. Additional phone checks are scheduled at the beginning of each 12 week part of the study. Participants will have a 50:50 chance of being on prazosin or placebo in the first 12 weeks of the study. For the second 12 weeks, all participants will take prazosin.

Study visits include a physical and neurological exam; memory testing; interviews with the caregiver about behaviors; and vital signs.

ELIGIBILITY:
Inclusion Criteria:

* No age limit
* Probable or Possible Alzheimer's Disease
* Disruptive agitated behaviors at least twice a week (overly anxious or excited, making offensive comments.....)
* Stable medications for 2 weeks
* Must have a caregiver who spends 10 hours per week caring for the participant and agrees to participate in all evaluation sessions

Exclusion Criteria:

* Cardiovascular: unstable angina, recent myocardial infarction, preexisting hypotension (systolic BP less than 110) or orthostatic hypotension (≥20 mmHg drop in systolic BP following 2 minutes of standing posture)
* Any unstable medical condition
* Exclusionary medications: current treatment with prazosin, other alpha-1 blockers (trazodone, sildenafil, vardenafil or tadalafil)
* Psychoactive medications: subjects may be psychoactive medication-free or be partial responders (by subjective assessment of referring health care professional) to one psychoactive medication from any of the following classes: antipsychotics, anticonvulsants, mood stabilizers, antidepressants, benzodiazepines, or buspirone. Partial response is defined as some improvement in agitated behavior but persistence of agitated behaviors severe enough to cause patient distress and/or difficulty with caregiving. Although not formally rated, this improvement is equivalent to a Clinical Global Impression of Change rating of no more than minimal improvement (improvement is noticed by not enough to improve patient function or caregiver's practical management of the patient).
* Psychiatric/behavioral: lifetime schizophrenia; current delirium, mania, depression, or uncontrolled persistent distressing psychotic symptoms (hallucinations, delusions), substance abuse, panic disorder, or any behavior which poses an immediate danger to patient or others or which results in the patient being too uncooperative to meet the requirements of study participation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elaine R Peskind, MD, Principal Investigator — University of Washington, VA Puget Sound Health Care System
Locations (1):
- Veterans Affairs Puget Sound Health Care System, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Period: Double Blind Phase
Arm/Group | Prazosin | Placebo
Started | 11 | 9
Completed | 7 | 7
Not Completed | 4 | 2
Period: Open-label Extension
Arm/Group | Prazosin | Placebo
Started | 5 (2 in the Prazosin arm of the Double Blind Phase elected not to enter the Open-Label extension) | 7
Completed | 4 | 6
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prazosin | Placebo | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 82.4 (10.5) | 78.7 (8.2) | 80.7 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 5 | 2 | 7
Total Neuropsychiatric Inventory score [Mean (Standard Deviation); unit: units on a scale] — The Neuropsychiatric Inventory is a scale that quantifies behavioral and psychiatric symptoms in patients with dementia. The scale ranges from 0 to 144, with 0 being no symptoms.
  units on a scale | 43.5 (16.2) | 40.9 (18.9) | 42.4 (17.1)
Brief Psychiatric Rating Scale [Mean (Standard Deviation); unit: units on a scale] — The Brief Psychiatric Rating Scale measures 18 psychiatric symptom domains. The scale ranges from 18 to 126, where 18 indicates no psychiatric symptoms.
  units on a scale | 45.4 (9.1) | 44.2 (9.5) | 44.9 (9.1)

OUTCOME MEASURES:

1. Primary Outcome: Alzheimer's Disease Cooperative Study - Clinical Global Impression of Change
Description: This scale represents the raters overall impression of improvement or worsening, and is assessed at the last visit. 1 = Marked improvement, 1 = Moderate improvement, 3 = Minimal improvement, 4 = No change, 5 = Minimal worsening, 6 = Moderate worsening, 7 = Marked worsening.
Time Frame: 12 Weeks after Baseline
Population: Any participant who had at least one follow-up assessment was included in the analysis. One participant in the Placebo group did not return for follow-up, and therefore was not included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prazosin | Placebo
Number analyzed (Participants) | 11 | 8
units on a scale | 2.5 (.25) | 2.43 (.28)

2. Secondary Outcome: Change in Brief Psychiatric Rating Scale Total Score
Description: Brief Psychiatric Rating Scale score change from Baseline to last observation. The Brief Psychiatric Rating Scale measures 18 psychiatric symptom domains. The scale ranges from 18 to 126, where 18 indicates no psychiatric symptoms.
Time Frame: 12 Weeks after Baseline
Population: One study participant in the Placebo group dropped out prior to first follow-up, although this subject is included in the statistical analysis to provide information on the outcome at baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prazosin | Placebo
Number analyzed (Participants) | 11 | 9
units on a scale | -9.8 (2.3) | -7.7 (2.8)

3. Primary Outcome: Change in Neuropsychiatric Inventory Score
Description: Neuropsychiatric Inventory score change from Baseline to last observation.The Neuropsychiatric Inventory is a scale that quantifies behavioral and psychiatric symptoms in patients with dementia. The scale ranges from 0 to 144, with 0 being no symptoms.
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prazosin | Placebo
Number analyzed (Participants) | 11 | 9
units on a scale | -23.4 (3.7) | -16.6 (4.5)

4. Secondary Outcome: Days in Study
Description: The number of days participants remained in the study during the Double Blind Phase. Please note that although the length of follow-up designated in the protocol was 12 weeks, a number of participants were in this phase longer (e.g. the dose titration phase took longer than 3 weeks, assessments were delayed due to scheduling conflicts, etc.) Therefore the length of time in the Double Blind Phase can exceed 12 weeks (84 days).
Time Frame: 12 weeks after Baseline
Population: 7 participants in the prazosin group were in the double-blind phase longer than 12 weeks (84 days). 4 participants in the placebo group were in the double-blind phase longer than 12 weeks (84 days).
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Prazosin | Placebo
Number analyzed (Participants) | 11 | 9
days | 87 (8) | 79 (9)

ADVERSE EVENTS:
Time Frame: 12 weeks.
Description: Known, common side effects for prazosin were specifically queried at each study visit.
Arm/Group | Prazosin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/9
Other Adverse Events (participants affected / at risk) | 11/11 | 9/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prazosin (N=11) | Placebo (N=9)
drowsiness (Nervous system disorders) | 7 (7) | 1 (1)
low energy (General disorders) | 4 (4) | 4 (4)
dizziness (General disorders) | 5 (5) | 1 (1)
lower extremity edema (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
headache (Nervous system disorders) | 3 (3) | 1 (1)
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
urinary tract infection (Renal and urinary disorders) | 1 (1) | 3 (3)
decreased appetite (General disorders) | 2 (2) | 1 (1)
nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
wound infection (Infections and infestations) | 0 (0) | 3 (3)
diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
gastrointestinal discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0)
increased agitation (Psychiatric disorders) | 0 (0) | 2 (2)
nocturnal enuresis (Renal and urinary disorders) | 2 (2) | 0 (0)
sleep disturbance (General disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No